CLINICAL TRIAL: NCT03854240
Title: Comparison of Ultrasound-Guided Classic And Lateral Approach Thoracolumbar Interfascial Plane Block For Pain Management Following Lumbar Laminectomy Surgery
Brief Title: Comparison of Ultrasound-Guided Classic And Lateral Approach Thoracolumbar Interfascial Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol University
Record Dates: First submitted 2019-02-23; First posted 2019-02-26 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Lumbar Disc Herniation
Keywords: Thoracolumbar Interfascial Plane Block; Pain Management; Lumbar Laminectomy Surgery
MeSH Terms: conditions — Intervertebral Disc Displacement; Agnosia | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Classic block (Group C) and modified block (Group M) will be performed following induction of general anesthesia, with patients in the prone position
Who Masked: Participant, Outcomes Assessor
Masking Description: the patient and the anesthesiologist who will evaluate postoperative pain will be blinded to the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic block (Group C) (Active Comparator): In group C, classic technique will be performed. US probe will be placed vertically at the L3 vertebrae level. After visualizing the hyperechoic shadow of the spinous process and interspinous muscles as an anatomical guide point, the probe will be moved forward to the lateral to visualize the longissimus and multifidus muscles. Between these muscles, block needle will be inserted within in plane technique in a lateral-to-medial direction in the interfascial plane. Once the needle tip will be placed within the interfacial plane and after careful aspiration to rule out intravascular needle placement, 2 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 20 mL will be injected in each side (total 40 mL)
  Interventions: Other: Classic block (Group C) and modified block (Group M) groups
- Modified block (Group M) (Active Comparator): In group M, modified technique will be performed. US probe will be placed vertically at the L3 vertebrae level. After visualizing the hyperechoic shadow of the spinous process and interspinous muscles as an anatomical guide point, the probe will be moved forward to the lateral to visualize the longissimus and iliocostal muscles. Between these muscles, block needle will be inserted within in plane technique in a medial-to-lateral direction in the interfascial plane. Once the needle tip will be placed within the interfacial plane and after careful aspiration to rule out intravascular needle placement, 2 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 20 mL will be injected in each side (total 40 mL)
  Interventions: Other: Classic block (Group C) and modified block (Group M) groups

INTERVENTIONS:
Other: Classic block (Group C) and modified block (Group M) groups — Classic block (Group C) and modified block (Group M) will be performed following induction of general anesthesia, with patients in the prone position by using ultrasound device

SUMMARY:
US-guided peripheral nerve blocks have been used increasingly due to the advantages of ultrasound in anesthesia practice. TLIP block is one of these nerve blocks performed under US guidance. In this technique, local anesthetic solution is injected between the multifidus and longissimus muscles nearly at the level of the 3rd lumbar vertebra and targets the dorsal rami of the thoracolumbar nerves. However, the visualisation of this technique may be difficult under ultrasound (US) guidance. Therefore, Ahiskalioglu et al. defined modified lateral technique of TLIP block as a new approach. The aim of this study is to compare US-guided classic and modified (lateral) techniques of TLIP block for postoperative analgesia management after lumbar laminectomy surgery .

DETAILED DESCRIPTION:
Spine surgery in thoracolumbar region is one of the most common surgeries performed for the treatment of leg and back pain 1. Pain management is especially important for these patients since chronic pain often occurs after surgery. Severe pain may occur at postoperative period in patients following lumbar disc herniation (LDH) operation. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced 1,2.

Regional anesthesia techniques may be preferred for postoperative analgesia management.Thoracolumbar interfascial plane (TLIP) block is a novel ultrasound guided regional analgesia technique.

Several techniques such as intravenous-intramuscular injections, and patient-controlled analgesia devices are usually performed for postoperative pain management. However, these methods may be ineffective in the pain treatment due to they are generally performed after pain has occurred. The analgesic agent may not reach a treatment concentration in the blood due to administrating doses intermittently 2.Opioids are one of the most preferred drugs among the analgesic agents. Parenteral opioids are generally performed for patients after surgery. However opioids have undesirable adverse events such as nausea, vomiting, itching, sedation and respiratory depression (opioid-related adverse events) 3.

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment. US-guided peripheral nerve blocks have been used increasingly due to the advantages of ultrasound in anesthesia practice. TLIP block is one of these nerve blocks performed under US guidance and defined by Hand et al. in 2015 2. In a retrospective study, it has been reported that this technique can provide effective analgesia after lumbar laminoplasty surgery by Ueshima et al 4. In this technique, local anesthetic solution is injected between the multifidus and longissimus muscles nearly at the level of the 3rd lumbar vertebra and targets the dorsal rami of the thoracolumbar nerves. However, the visualisation of this technique may be difficult under ultrasound (US) guidance. Therefore, Ahiskalioglu et al. defined modified lateral technique of TLIP block as a new approach 5. Ahiskalioglu et al. have reported that this approach has some advantages. Firstly, sonographic visualisation is more easily than the classical technique. Secondly, insertion of the needle from medial to lateral direction reduces the risk of possible neuraxial injection 5.

The aim of this study is to compare US-guided classic and modified (lateral) techniques of TLIP block for postoperative analgesia management after lumbar laminectomy surgery . The primary aim is to compare perioperative and postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting) and complications due to blocks.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* scheduled for lumbar laminectomy surgery

Exclusion Criteria:

* bleeding diathesis
* receiving anticoagulant treatment
* known local anesthetics and opioid allergy
* infection of the skin at the site of the needle puncture
* pregnancy or lactation
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
opioid consumption | up to 3 months
  The primary aim is to compare perioperative and postoperative opioid consumption

SECONDARY OUTCOMES:
Visual analogue scores (VAS) | up to 3 months
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not share IPD

REFERENCES:
- [Background] Ahiskalioglu A, Alici HA, Selvitopi K, Yayik AM. Ultrasonography-guided modified thoracolumbar interfascial plane block: a new approach. Can J Anaesth. 2017 Jul;64(7):775-776. doi: 10.1007/s12630-017-0851-y. Epub 2017 Feb 27. No abstract available. PMID 28243853
- [Background] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600
- [Background] Ueshima H, Ozawa T, Toyone T, Otake H. Efficacy of the Thoracolumbar Interfascial Plane Block for Lumbar Laminoplasty: A Retrospective Study. Asian Spine J. 2017 Oct;11(5):722-725. doi: 10.4184/asj.2017.11.5.722. Epub 2017 Oct 11. PMID 29093781